CLINICAL TRIAL: NCT03947086
Title: Transcranial Direct Current Stimulation for Cognitive Rehabilitation of Children With Autistic Spectrum Disorders
Brief Title: Neurostimulation for Cognitive Rehabilitation in Autistic Spectrum Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Jéssica Bruna Santana Silva, Principal Investigator, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1221-6178
Record Dates: First submitted 2019-04-30; First posted 2019-05-13 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Autistic Disorders Spectrum
Keywords: Autistic disorder; Neuromodulation; Social cognition; Executive functions; Eye tracking
MeSH Terms: conditions — Child Development Disorders, Pervasive; Autistic Disorder | interventions — Transcranial Direct Current Stimulation; Cognitive Training

STUDY DESIGN:
Intervention Model Description: this study is a sham-controlled, double-blind, randomized clinical trial aiming to evaluate the efficacy of anodic TDCS in aspects of social cognition of children between 8 and 12 years old with mild ASD. In total there will be 16 children, diagnosed with ASD according DSM-V, will be randomized to two groups, one with active stimulation (1.5 mA) and the other with a placebo current, in which the anode will be positioned over the left dorsolateral prefrontal cortex (F3), while the cathode (reference electrode) will be placed in the right supraorbital area. The intervention will be applied for 5 consecutive days for 20 minutes. Participants and investigators will be blinded. Furthermore, everyone will receive Social Cognition Training concomitantly with neurostimulation to enhance social skills in children with ASD. Patients will undergo three social cognitive assessments: at baseline, week 2 (after stimulation), and 1 month later (follow up).
Who Masked: Participant, Investigator
Masking Description: Participants enrolled in the study using the eligibility criteria will be allocated randomly, with 1: 1 block exchange. A random number generator will be used through an online randomization program (www.random.org). Hidden allocation will be employed with numbered, opaque and sealed sequential envelopes, so that the person in charge of the allocation will not have contact with the patients, nor with the work of the others.
  In addition, all examiners will be blind as to the type of treatment the patient will receive (active stimulation or sham-controlled), which will be done by a specific investigator. The protocol for simulated current is identical, but the device ceases to emit current after 30 seconds of initiation of pacing. In this way, the effects of the active stimulation by short stimulation period are simulated, without inducing clinical effects. These factors characterize this trial as a double-blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active TDCS Group (Active Comparator): Participants will receive active Transcranial Direct Current Stimulation (TDCS) (1.5 mA). Furthermore, everyone will receive Social Cognition Training concomitantly with neurostimulation to enhance social skills.
  Interventions: Device: Transcranial Direct Current Stimulation (TDCS)- Active; Behavioral: Cognitive Training
- Sham tDCS Group (Sham Comparator): Participants will receive sham TDCS. The protocol is identical for placebo stimulation, but the current will stop after 30 seconds from the start of stimulation. Furthermore, everyone will receive Social Cognition Training concomitantly with neurostimulation to enhance social skills.
  Interventions: Device: Transcranial Direct Current Stimulation (TDCS)- Sham; Behavioral: Cognitive Training

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (TDCS)- Active — A constant current stimulator (TCT Research Limited) will be used using electrodes of 5 × 5 cm2 embedded in saline (0.9 % NaCl) and application of 1.5 mA current for 20 minutes for 5 consecutive days. The cathode will be positioned in the right supra-orbital region, and while the anode will have the following provision in the left dorsolateral prefrontal cortex (F3).
  Arms: Active TDCS Group
Device: Transcranial Direct Current Stimulation (TDCS)- Sham — The protocol for participants receiving simulated current is identical, but the device ceases to emit current after 30 seconds of initiation of pacing.
  Arms: Sham tDCS Group
Behavioral: Cognitive Training — Considering that the effects of TDCS are potentiated when applied during the execution of a task (online) (Miniussi, & Ruzzoli, 2013), in the present study all participants received cognitive training, performed concomitantly with neurostimulation.
  Cognitive training consists of two parts: standardized tasks directed to social cognition and activities that stimulate executive functions. The first part consists of tasks contained in a battery of social games (Gao & Maurer, 2009; Dillon, Kannan, Dean, Spelke, & Duflo, 2017). While the tasks directed to the executive domain are, namely: running mazes, assembling figures, completing parts of figures and the Super Lynx Memory Game. All participants, regardless of whether they underwent active or simulated stimulation, received cognitive training, respecting the ethical principles of ensuring therapeutic assistance to those involved.

SUMMARY:
This study is a clinical trial aims investigate the effects of neurostimulation in the treatment of children with mild ASD, specifically the action of tDCS on social cognition skills. tDCS can modulate neuronal activity in patients with ASD. Specifically, this technique has shown to be a promising tool in the promotion of social neuroplasticity, aiming at more adaptive social interactions. In this sense, it was hypothesized that participants treated with active tDCS will present better performance in social cognition tests than those submitted to sessions with simulated current.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a neurodevelopmental disorder that has multiple causes and very heterogeneous degrees. The main symptoms involve deficits in social interactions, difficulties in verbal and nonverbal communication, repetitive and stereotyped movements, and restricted patterns of interest. In the context of ASD rehabilitation, there is no specific treatment for autism so far, being the behavioral therapy the most used therapeutic strategy, but with still unsatisfactory results. Transcranial Direct Current Stimulation (tDCS) has been shown to be a promising technique for the treatment of different disorders, including ASD. The tDCS consists of electrical signals emitted through two electrodes in different areas of the scalp, according to the purpose of the study. The anodic current reduces the firing threshold of the neurons that are located in the cortex (that is, they increase the spontaneous firing of these neurons), whereas the cathodic current increases the firing threshold of the neurons (that is, it inhibits the activity of these neurons). Considering neuroplasticity mechanisms as fundamental in cognitive processing, tDCS becomes a promising tool in neuropsychological rehabilitation in the treatment of autistic symptoms. Previous research using protomagnetic resonance spectroscopy (H-MRS) showed lower levels of N-acetyl aspartate (NAA, a marker of mitochondrial function and neuronal density) in the left DLFPC (F3) of autistic patients, compared to healthy individuals. The findings suggest that left DLFPC dysfunction may be a component of the pathogenesis of autism. Such aspects could explain why anodic neurostimulation in F3 can improve the efficacy of autism treatment through the beneficial effects on the cognitive processes associated with DLFPC activity, such as attention and memory, executive functions, and social cognition. Social cognition can be understood as a neurobiological process that facilitates the interpretation of social signs, leading individuals to behave adaptively. In this perspective, investigations have been made that use noninvasive neuromodulatory techniques as promising tools for the promotion of social neuroplasticity, that is, the modulation of the functional and structural substrates of the nervous system associated with social cognition aiming at more adaptive social interactions.In this sense, this study is a sham-controlled, double-blind, randomized clinical trial aiming to evaluate the efficacy of anodic tDCS in aspects of social cognition of children with mild ASD. Considering that tDCS can modulate neuronal activity in patients with ASD, presented as a promising tool in the promotion of social neuroplasticity, it was hypothesized that participants treated with active current will present better performance in the social cognition tests than those submitted to sessions with simulated current. Participants treated with active current will present less number and duration of fixations in the ocular tracing during the execution of the test of recognition of emotional expressions than those submitted to the sessions with simulated current. Furthermore, cognitive processes such as executive functions are essential for social cognition because they enable the individual to engage in socially relevant activities, make decisions and behaviors to achieve goals. Deficits in social cognition as well as executive functioning have been considered central elements in the understanding and functionality of people with ASD. Thus, it was hypothesized that participants who are treated with active current will present better performance in the tests of executive functions than those submitted to the sessions with simulated current. Participants treated with active current will present less number and duration of fixations during ocular screening in the executive function test than those submitted to the simulated current sessions. Considering that there were no prior data on the effects of tDCS on patients with ASD using the primary outcome measure of the present study, a formal sample size calculation was not possible; thus, it was estimated that enrolling 20 patients would be a reasonable approach for an exploratory trial. Patients are being recruited from the appointment of rehabilitators of multidisciplinary rehabilitation centers for temporary or permanent disability and global developmental disorders in Paraíba, Brazil. Children diagnosed with ASD according DSM-V, will be randomized to two groups, one with active stimulation (1.5 mA) and the other with a sham current, in which the anode will be positioned over the left dorsolateral prefrontal cortex (F3), while the cathode (reference electrode) will be placed in the right supraorbital area. The intervention will be applied for 5 consecutive days for 20 minutes. Furthermore, everyone will receive Social Cognition Training concomitantly with neurostimulation to enhance social skills in children with ASD. To control adverse effects, reports of patients with feelings/sensations of itching, tingling, burning, headache or other discomfort (1 none, 2 mild, 3 moderate, or 4 strong) will be recorded, along with whether this effect could be related to stimulation on a Likert scale; 1 (no relation) to 5 (strongly related).

The Descriptive and inferential statistical analyzes will be performed through SPSS (Statistical package for the social sciences), version 20. The design of the statistical analyzes is based on previous literature studies of randomized and placebo-controlled clinical trials using tDCS. The intention-to-treat analysis will be used with the last observation carried forward method for patients who initiate treatment and receive at least 1 session. In this way, all participants, including in case of withdrawal of the treatment before its completion, will be included in the analysis. It will be used as significance level p <0.05.

The descriptive statistics will be used to describe the clinical and sociodemographic characteristics, as well as the primary and secondary outcomes of each group in T0. The groups will be compared using Student's t test for continuous variables, or chi-square, for categorical variables.

The evaluation and efficacy of tDCS in all variables of the primary and secondary outcomes will be examined with mixed two-way ANOVA, repeated measures, one dependent variable and two independent variables, one intra-group (time, with 3 levels, T0, T2 and T3), and between-groups (two levels: Active, Sham). Covariance analyzes (ANCOVA) will be used to identify significant differences between groups using the T0 scores as covariables. In addition, adverse effects will be analyzed using the chi-square test.

Linear logistic regression will be used to identify predictors of response. The independent variables are: tDCS active and sham, the predictive variables, analyzed one at a time, will be: age and severity of symptoms. Patients will undergo three social cognitive assessments: at baseline, week 2 (after stimulation), and 1 month later. Adverse effects will be computed at each session. Thus, this clinical trial aims to investigate the combined effects of transcranial direct current stimulation and social cognition training in improving the social skills of children with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ASD
* Degree of mild autistic symptomatology
* Normal or corrected acuity.

Exclusion Criteria:

* Intellectual deficits
* Cardiac pacemaker or implanted metallic or electronic device
* Severe neurological disorders
* Poor skull formation
* Epilepsy

Ages: 8 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2018-04-30 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
Facial emotion recognition | The test will be measured immediately before the intervention.
  Images of facial expressions of emotion of children of diverse ethnicities will be presented. We used 20 images of emotional expressions of the test of emotional knowledge elaborated by Izard, Hankins, Schultz, Tentracosta and King (2003). The following emotional faces of both sexes will be used: happy, sad, angry, fear / surprised and neutral, presented at random and for 4 seconds each. During the recognition of the emotional expressions, the 300 Hz binocular Eye Tracker Tobii was used to monitor eye movements.
  .
Facial emotion recognition | The test will be measured immediately after the intervention.
  Images of facial expressions of emotion of children of diverse ethnicities will be presented. We used 20 images of emotional expressions of the test of emotional knowledge elaborated by Izard, Hankins, Schultz, Tentracosta and King (2003). The following emotional faces of both sexes will be used: happy, sad, angry, fear / surprised and neutral, presented at random and for 4 seconds each. During the recognition of the emotional expressions, the 300 Hz binocular Eye Tracker Tobii was used to monitor eye movements.
  .
Facial emotion recognition | The test will be measured 4 weeks after the intervention.
  Images of facial expressions of emotion of children of diverse ethnicities will be presented. We used 20 images of emotional expressions of the test of emotional knowledge elaborated by Izard, Hankins, Schultz, Tentracosta and King. The following emotional faces of both sexes will be used: happy, sad, angry, fear / surprised and neutral, presented at random and for 4 seconds each. During the recognition of the emotional expressions, the 300 Hz binocular Eye Tracker Tobii was used to monitor eye movements.
  .
Theory of mind- Verbal task | The test will be measured immediately before the intervention.
  The subtest theory of mind contained in Nepsy II neuropsychological battery will be used. The test includes two tasks: the verbal task evaluates the understanding and perception of self-intention and of the other, deception, beliefs, pretending, and imitation through stories, figures, and questions. The contextual task evaluates the ability to relate a situation to emotion in a specific social context.
Theory of mind- Contextual task | The test will be measured immediately before the intervention.
  The subtest theory of mind contained in Nepsy II neuropsychological battery will be used. The test includes two tasks: the verbal task evaluates the understanding and perception of self-intention and of the other, deception, beliefs, pretending, and imitation through stories, figures, and questions. The contextual task evaluates the ability to relate a situation to emotion in a specific social context.
Theory of mind- Verbal task | The test will be measured immediately after the intervention.
  The subtest theory of mind contained in Nepsy II neuropsychological battery will be used. The test includes two tasks: the verbal task evaluates the understanding and perception of self-intention and of the other, deception, beliefs, pretending, and imitation through stories, figures, and questions. The contextual task evaluates the ability to relate a situation to emotion in a specific social context.
Theory of mind- Contextual task | The test will be measured immediately after the intervention.
  The subtest theory of mind contained in Nepsy II neuropsychological battery will be used. The test includes two tasks: the verbal task evaluates the understanding and perception of self-intention and of the other, deception, beliefs, pretending, and imitation through stories, figures, and questions. The contextual task evaluates the ability to relate a situation to emotion in a specific social context.
Theory of mind- Verbal task | The test will be measured 4 weeks after the intervention.
  The subtest theory of mind contained in Nepsy II neuropsychological battery will be used. The test includes two tasks: the verbal task evaluates the understanding and perception of self-intention and of the other, deception, beliefs, pretending, and imitation through stories, figures, and questions. The contextual task evaluates the ability to relate a situation to emotion in a specific social context.
Theory of mind- Contextual task | The test will be measured 4 weeks after the intervention.
  The subtest theory of mind contained in Nepsy II neuropsychological battery will be used. The test includes two tasks: the verbal task evaluates the understanding and perception of self-intention and of the other, deception, beliefs, pretending, and imitation through stories, figures, and questions. The contextual task evaluates the ability to relate a situation to emotion in a specific social context.

SECONDARY OUTCOMES:
Memory for Digit Span | The test will be measured immediately before the intervention.
  The measure was used to evaluate the operational memory. There are two parts to the Memory for Digit Span assessment: Digits Forward and Digits Backward. Each tap distinct but interdependent cognitive functions. Digits Forward primarily taps short-term auditory memory while Digits Backward measures the child's ability to manipulate verbal information while in temporary storage. In Digits Forward, the child listens to and repeats a sequence of numbers spoken aloud by the interviewer. In Digits Backward, the child listens to a sequence of numbers and repeats them in reverse order.
Memory for Digit Span | The test will be measured immediately after the intervention.
  The measure was used to evaluate the operational memory. There are two parts to the Memory for Digit Span assessment: Digits Forward and Digits Backward. Each tap distinct but interdependent cognitive functions. Digits Forward primarily taps short-term auditory memory while Digits Backward measures the child's ability to manipulate verbal information while in temporary storage. In Digits Forward, the child listens to and repeats a sequence of numbers spoken aloud by the interviewer. In Digits Backward, the child listens to a sequence of numbers and repeats them in reverse order.
Memory for Digit Span | The test will be measured 4 weeks after the intervention.
  The measure was used to evaluate the operational memory. There are two parts to the Memory for Digit Span assessment: Digits Forward and Digits Backward. Each tap distinct but interdependent cognitive functions. Digits Forward primarily taps short-term auditory memory while Digits Backward measures the child's ability to manipulate verbal information while in temporary storage. In Digits Forward, the child listens to and repeats a sequence of numbers spoken aloud by the interviewer. In Digits Backward, the child listens to a sequence of numbers and repeats them in reverse order.
Trail Making Test A e B | The test will be measured immediately before the intervention.
  The TMT measures attention, speed, and mental flexibility. Part A requires the individual to draw lines to connect 25 encircled numbers distributed on a page. Part A tests visual scanning, numeric sequencing, and visuomotor speed. Part B is similar except the person must alternate between numbers and letters and is believed to be more difficult and takes longer to complete. Part B tests cognitive demands including visual motor and visual spatial abilities and mental flexibility.
Trail Making Test A e B | The test will be measured immediately after the intervention.
  The TMT measures attention, speed, and mental flexibility. Part A requires the individual to draw lines to connect 25 encircled numbers distributed on a page. Part A tests visual scanning, numeric sequencing, and visuomotor speed. Part B is similar except the person must alternate between numbers and letters and is believed to be more difficult and takes longer to complete. Part B tests cognitive demands including visual motor and visual spatial abilities and mental flexibility.
Trail Making Test A e B | The test will be measured 4 weeks after the intervention.
  The TMT measures attention, speed, and mental flexibility. Part A requires the individual to draw lines to connect 25 encircled numbers distributed on a page. Part A tests visual scanning, numeric sequencing, and visuomotor speed. Part B is similar except the person must alternate between numbers and letters and is believed to be more difficult and takes longer to complete. Part B tests cognitive demands including visual motor and visual spatial abilities and mental flexibility.
Seven Errors Test | The test will be measured immediately before the intervention.
  This test aims to evaluate executive functions globally. The test consists of two different pairs of figures: a pair of figures of one elephant, and another pair refers to a boat. Each pair has the original figure and the figure containing the errors, both appear simultaneously on the screen, side by side, and the participant must identify the errors / differences between the figures. The 300 Hz binocular Eye Tracker Tobii was used to monitor eye movements during the test.
Seven Errors Test | The test will be measured immediately after the intervention.
  This test aims to evaluate executive functions globally. The test consists of two different pairs of figures: a pair of figures of one elephant, and another pair refers to a boat. Each pair has the original figure and the figure containing the errors, both appear simultaneously on the screen, side by side, and the participant must identify the errors / differences between the figures. The 300 Hz binocular Eye Tracker Tobii was used to monitor eye movements during the test.
Seven Errors Test | The test will be measured 4 weeks after the intervention.
  This test aims to evaluate executive functions globally. The test consists of two different pairs of figures: a pair of figures of one elephant, and another pair refers to a boat. Each pair has the original figure and the figure containing the errors, both appear simultaneously on the screen, side by side, and the participant must identify the errors / differences between the figures. The 300 Hz binocular Eye Tracker Tobii was used to monitor eye movements during the test.

CONTACTS AND LOCATIONS:
Overall Officials: Jéssica B Santana, Master, Principal Investigator — Federal University of Paraíba; Natanael A Santos, PhD, Study Director — Federal University of Paraíba
Locations (1):
- Gabriela Medeiros, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amatachaya A, Auvichayapat N, Patjanasoontorn N, Suphakunpinyo C, Ngernyam N, Aree-Uea B, Keeratitanont K, Auvichayapat P. Effect of anodal transcranial direct current stimulation on autism: a randomized double-blind crossover trial. Behav Neurol. 2014;2014:173073. doi: 10.1155/2014/173073. Epub 2014 Oct 30. PMID 25530675
- [Background] Amatachaya A, Jensen MP, Patjanasoontorn N, Auvichayapat N, Suphakunpinyo C, Janjarasjitt S, Ngernyam N, Aree-uea B, Auvichayapat P. The short-term effects of transcranial direct current stimulation on electroencephalography in children with autism: a randomized crossover controlled trial. Behav Neurol. 2015;2015:928631. doi: 10.1155/2015/928631. Epub 2015 Mar 12. PMID 25861158
- [Background] Jamil A, Batsikadze G, Kuo HI, Labruna L, Hasan A, Paulus W, Nitsche MA. Systematic evaluation of the impact of stimulation intensity on neuroplastic after-effects induced by transcranial direct current stimulation. J Physiol. 2017 Feb 15;595(4):1273-1288. doi: 10.1113/JP272738. Epub 2016 Nov 8. PMID 27723104
- [Background] Boggio PS, Asthana MK, Costa TL, Valasek CA, Osorio AA. Promoting social plasticity in developmental disorders with non-invasive brain stimulation techniques. Front Neurosci. 2015 Sep 1;9:294. doi: 10.3389/fnins.2015.00294. eCollection 2015. PMID 26388712
- [Background] Brunoni AR, Nitsche MA, Bolognini N, Bikson M, Wagner T, Merabet L, Edwards DJ, Valero-Cabre A, Rotenberg A, Pascual-Leone A, Ferrucci R, Priori A, Boggio PS, Fregni F. Clinical research with transcranial direct current stimulation (tDCS): challenges and future directions. Brain Stimul. 2012 Jul;5(3):175-195. doi: 10.1016/j.brs.2011.03.002. Epub 2011 Apr 1. PMID 22037126
- [Background] Couture SM, Penn DL, Roberts DL. The functional significance of social cognition in schizophrenia: a review. Schizophr Bull. 2006 Oct;32 Suppl 1(Suppl 1):S44-63. doi: 10.1093/schbul/sbl029. Epub 2006 Aug 17. PMID 16916889
- [Background] Demirtas-Tatlidede A, Vahabzadeh-Hagh AM, Pascual-Leone A. Can noninvasive brain stimulation enhance cognition in neuropsychiatric disorders? Neuropharmacology. 2013 Jan;64:566-78. doi: 10.1016/j.neuropharm.2012.06.020. Epub 2012 Jun 28. PMID 22749945
- [Background] Dillon MR, Kannan H, Dean JT, Spelke ES, Duflo E. Cognitive science in the field: A preschool intervention durably enhances intuitive but not formal mathematics. Science. 2017 Jul 7;357(6346):47-55. doi: 10.1126/science.aal4724. PMID 28684518
- [Background] Gao X, Maurer D. Influence of intensity on children's sensitivity to happy, sad, and fearful facial expressions. J Exp Child Psychol. 2009 Apr;102(4):503-21. doi: 10.1016/j.jecp.2008.11.002. Epub 2009 Jan 4. PMID 19124135
- [Background] Kucharska-Pietura K, Mortimer A. Can antipsychotics improve social cognition in patients with schizophrenia? CNS Drugs. 2013 May;27(5):335-43. doi: 10.1007/s40263-013-0047-0. PMID 23533009
- [Background] Kuo MF, Paulus W, Nitsche MA. Therapeutic effects of non-invasive brain stimulation with direct currents (tDCS) in neuropsychiatric diseases. Neuroimage. 2014 Jan 15;85 Pt 3:948-60. doi: 10.1016/j.neuroimage.2013.05.117. Epub 2013 Jun 4. PMID 23747962
- [Background] Nitsche MA, Cohen LG, Wassermann EM, Priori A, Lang N, Antal A, Paulus W, Hummel F, Boggio PS, Fregni F, Pascual-Leone A. Transcranial direct current stimulation: State of the art 2008. Brain Stimul. 2008 Jul;1(3):206-23. doi: 10.1016/j.brs.2008.06.004. Epub 2008 Jul 1. PMID 20633386
- [Background] Muszkat D, Polanczyk GV, Dias TG, Brunoni AR. Transcranial Direct Current Stimulation in Child and Adolescent Psychiatry. J Child Adolesc Psychopharmacol. 2016 Sep;26(7):590-7. doi: 10.1089/cap.2015.0172. Epub 2016 Mar 30. PMID 27027666